CLINICAL TRIAL: NCT04401111
Title: Multiparametric Evaluation of One-year Outcomes in Survivors of the Severe COVID-19 Pneumonia After Intensive Care Unit
Brief Title: One-year Outcomes in Survivors of the Severe COVID-19 Pneumonia (CO-Qo-ICU)
Acronym: CO-Qo-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20reamedcovid04
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: COVID; ARDS; Quality of Life
Keywords: Long term prognosis; Six-minute walk test; Restrictive syndrom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivors of Intensive care unit patients: Survivors of severe COVID-19 pneumonia after intensive care unit

SUMMARY:
Many of the patients hospitalized for a severe form of SARSCoV-2 respiratory impairment require prolonged intensive care that can be complicated in the short term, In the medium and long term, physical and psychological sequelae can affect patients' quality of life and prevent a return to normal working life.

To date, there is little data on the fate of patients treated in Resuscitation for a severe form of COVID-19, both in terms of respiratory sequelae, as well as in terms of psychological sequelae and their quality of life. The objective of this study is to be able to describe and evaluate the possible physical and psychological sequelae and quality of life of patients hospitalized in Resuscitation for a severe form of COVID-19 in the short (3 and 6 months), medium (1 year) and long (5 years) End of their stay in ICU. To do this, we want to carry out a prospective, observational and monocentric study in the consultation department of the Nice CHU. All patients admitted to Resuscitation for a severe form of COVID-19 who have accepted the longitudinal medical follow-up proposed by the Nice CHU will be included in the study and data from the computerized medical record will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in ICU for an ARDS table
* PCR SARSCoV-2 nasopharyngeal or positive pulmonary samples

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated for COVID-19 in Intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment at 3 months of stay in ICU patients hospitalized for a severe form of COVID-19 | 5 years
  SF-36 score calculation at 3 months of inpatient ICU stay for severe COVID-19

SECONDARY OUTCOMES:
Quality of Life Assessment at 6 months, 1 year and 5 years of Inpatient Resuscitation for severe COVID-19 | 5 years
  Quality of Life Assessment at 6 months, 1 year and 5 years of Inpatient Resuscitation for severe COVID-19
Assessment of respiratory function and lung lesions at 3 months, 6 months, 1 year and 5 years of hospitalized patients in ICU for severe COVID-19. | 5 years
  Vital and total lung capacity measurement when performing respiratory functional scans
Stress-based assessment of respiratory function at 3 months, 6 months, 1 year and 5 years of hospitalized ICU for severe COVID-19 | 5 years
  Measurement of the extent of pulmonary parenchymal lesions when performing a chest CT scan at 3 months, 6 months, 1 year and 5 years of hospitalized patients in ICU for severe COVID-19
Assessment of resuscitation neuromyopathy at 3 months, 6 months, 1 year and 5 years of hospitalized patients in Resuscitation for severe COVID-19 | 5 years
  Measurement of CKD score at 3 months, 6 months, 1 year and 5 years of hospitalized patient ICU for severe COVID-19. This score described in Appendix 2 is the recommended score for assessing resuscitation neuromyopathy
Left and Right Cardiac Function Assessment at 3 months, 6 months, 1 year and 5 years of Inpatient Resuscitation for severe COVID-19 | 5 years
  Measurement of left and right ventricular ejection fraction when performing a transthoracic cardiac ultrasound at 3 months, 6 months, 1 year and 5 years of hospitalized ICU for a severe form of COVID-19
Psychological evaluation at 3 months, 6 months, 1 year and 5 years of stay in Intensive Care for patients hospitalized for a serious form of COVID-19 | 5 years
  Evaluation des scores IES-R (Impact of Event Scale Revised) et HAD (Hospital Anxiety and Depression scale)
Evaluation of the possible impact on professional activity at 3 months, 6 months, 1 year and 5 years of stay in Intensive Care for patients hospitalized for a serious form of COVID-19 | 5 years
  Measure the return to work rate (full-time, half-time, <half-time, none) at 3 months, 6 months, 1 year and 5 years of hospitalized Resuscitation for severe COVID-19.
Assessment of the 3-month, 6-month, 1-year and 5-year hospitalization rate for hospitalized patients with severe COVID-19. | 5 years
  The number of hospitalizations and the number of days spent in hospital at 3 months, 6 months, 1 year and 5 years of hospitalized patients in ICU for severe COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
No Data sharing plan has been established